CLINICAL TRIAL: NCT06414577
Title: A Single-Arm Phase II Clinical Study of Irinotecan Liposomes in Combination With Nituzumab for the Treatment of Recurrent/Metastatic Nasopharyngeal Carcinoma After Failure of First-Line or Higher Immunotherapy
Brief Title: Irinotecan Liposomes in Combination With Nituzumab for the Treatment of Recurrent/Metastatic Nasopharyngeal Carcinoma After Failure of First-Line or Higher Immunotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: XIANG YANQUN (Other)
Responsible Party: Sponsor-Investigator, XIANG YANQUN, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-110-01
Record Dates: First submitted 2024-04-29; First posted 2024-05-16 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: liposomal irinotecan administered intravenously at a dose of 70 mg/m2 on day 1, along with nituzumab given at a dose of 400 mg via intravenous injection on the same day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan Liposomes combined With Nituzumab (Experimental)
  Interventions: Drug: Irinotecan Liposomal combined With Nituzumab

INTERVENTIONS:
Drug: Irinotecan Liposomal combined With Nituzumab — Irinotecan liposomal: 70mg/m2, ivgtt, d1; Nituzumab: 400 mg, igvtt, d1 One treatment cycle every two weeks for up to 8 cycles, or until disease progression, intolerable toxicity, death, and investigator judgment of no further benefit

SUMMARY:
Nasopharyngeal cancer is a malignant tumor that arises from the cells of the nasopharyngeal epithelium, with its occurrence spread across different regions worldwide. Recent data from China in 2015 revealed approximately 6.0 million new cases of nasopharyngeal cancer, leading to approximately 34,000 deaths. When choosing a chemotherapy regimen for patients with metastatic nasopharyngeal cancer, the gemcitabine and cisplatin combination (GP) is typically recommended as the initial treatment. However, it is common for patients to experience disease progression after receiving first-line chemotherapy, highlighting the importance of a well-defined second-line treatment plan.

Recent clinical studies have indicated that combining nituzumab with radiotherapy can enhance treatment efficacy with minimal side effects, providing promising results for advanced nasopharyngeal cancer patients. Additionally, the use of irinotecan liposome injection has proved beneficial in modifying the drug's pharmacokinetics, resulting in improved drug delivery to the tumor site while reducing toxicity in healthy tissues. This study aims to explore the effectiveness and safety of combining irinotecan liposome with nituzumab treatment for recurrent metastatic nasopharyngeal carcinoma that has not responded to initial immunotherapy.

Participants selected for this clinical trial will receive a treatment regimen consisting of liposomal irinotecan administered intravenously at a dose of 70 mg/m2 on day 1, along with nituzumab given at a dose of 400 mg via intravenous injection on the same day. This treatment cycle will be repeated every two weeks for a maximum of eight cycles, or until disease progression, intolerable side effects, or other criteria necessitating discontinuation of treatment as determined by the investigator. By evaluating the efficacy and safety of this combined regimen, investigators aim to establish a novel therapeutic approach for managing advanced nasopharyngeal carcinoma in the context of current immunotherapy advancements.

ELIGIBILITY:
Inclusion Criteria:

* 1. subjects volunteered to participate in the study and signed an informed consent form (ICF); 2. age ≥ 18 years; and 3. previous histopathological diagnosis of non-keratinizing carcinoma of the nasopharynx (differentiated or undifferentiated, i.e., WHO classification type II or III); and 4. positive EGFR test; 5. patients with recurrent/metastatic nasopharyngeal cancer who have received prior treatment with first-line or higher standard regimens containing PD-1/PD-L1 inhibitors; 6. at least 1 evaluable lesion at baseline according to RECIST 1.1 criteria; the area must not have received prior radiotherapy or there must be evidence of significant progression of the lesion after completion of radiotherapy; 7. ECOG score 0 to 1; expected survival ≥ 3 months 8. No serious cardiac, pulmonary, hepatic, renal or other vital organ dysfunction; normal hepatic and renal function: AST, ALT <2.5 times the upper limit of normal, total bilirubin <1.5 times the upper limit of normal; serum creatinine ≤1.5 × the upper limit of normal and creatinine clearance ≥ 30 mL/min; adequate bone marrow function: peripheral blood leukocytes >4.0 × 109/L, neutrophils >1.0 × 109/L, hemoglobin >90%. 109/L, hemoglobin > 90 g/L, platelets > 100 × 109/L;

Exclusion Criteria:

* 1. history of hypersensitivity to monoclonal antibodies; hypersensitivity to liposomal irinotecan; 2. use of a strong inducer of CYP3A4 within 2 weeks or a strong inhibitor of CYP3A4 or a strong inhibitor of UGT1A1 within 1 week prior to the first administration of the trial drug; 3. expected survival time < 3 months; 4. active hepatitis B (HbsAg or HBcAb positive and HBV DNA ≥ 2000 IU/mL), active hepatitis C (HCV antibody positive and HCVRNA above the lower limit of the study center's assay); if the patient has normal liver function and is taking concomitant antiviral medication, eligibility for enrollment will be determined by the investigator; 5. patients who are HIV antibody positive; and 6. active bacterial, fungal, viral, or interstitial pneumonia requiring systemic therapy within 1 week prior to the first dose of study drug; and 7. have received antineoplastic therapy such as chemotherapy, small molecule inhibitors, immunotherapy (e.g., interleukin, interferon, or thymosin) within 4 weeks or 5 half-lives, whichever is shorter, but at least 2 weeks prior to the first dose of study drug; 8. treatment with a proprietary Chinese medicine with antitumor activity within 14 days prior to administration; treatment with another clinically investigational drug within 4 weeks prior to the first dose; 9. has undergone major surgery within 3 months prior to the first dose, or plans to undergo major surgery during the study period 10. has had a serious embolic event, e.g., cerebrovascular accident (including transient ischemic attack), pulmonary embolism, within 6 months prior to screening; 11. active malignancy within 2 years prior to the first study drug administration, with the exception of nasopharyngeal carcinoma, which is being studied in this trial, and any locally curable tumors that have undergone radical therapy (e.g., resected basal or squamous cell skin cancer, superficial bladder cardiac abnormalities including: carcinoma of the bladder, carcinoma of the cervix, or breast carcinoma in situ) 12. severe cardiovascular disease within 6 months prior to enrollment, including but not limited to the following:

  * Acute myocardial infarction, unstable angina, coronary angioplasty or stenting, deep vein thrombosis, stroke; ② New York Heart Association class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) <50%; ③ Abnormal electrocardiograms (ECGs) of clinical significance at the time of screening, as assessed by the investigator; 13. women who are pregnant or breastfeeding; 14. any serious and/or uncontrollable medical condition, as determined by the investigator, other medical conditions that may interfere with the patient's participation in this study (including, but not limited to, uncontrolled diabetes mellitus, renal disease requiring dialysis, severe liver disease, life-threatening autoimmune and bleeding disorders, substance abuse, neurological disorders, etc.);; and 15. other conditions judged by the investigator to be unsuitable for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-03-23 (Estimated); Study Completion 2025-03-23 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | up to 2 years

SECONDARY OUTCOMES:
one-year overall survival(OS) rate | up to 2 years
one-year progression-free survival(PFS) rate | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No